CLINICAL TRIAL: NCT04180254
Title: Evaluation and Optimization of Hearing Devices in 3-D Complex Audio Environments Study 3
Brief Title: Evaluation and Optimization of Hearing Devices in 3-D Complex Audio Environments Study 3 (HEAR3D_CE3)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sonova AG (Industry)
Collaborators: Swiss Commission for Technology and Innovation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2017-02051-3
Record Dates: First submitted 2019-11-25; First posted 2019-11-27 (Actual); Last update posted 2020-09-02 (Actual); Status verified 2020-09

CONDITIONS: Ability, Spatial
MeSH Terms: conditions — Spatial Navigation

STUDY DESIGN:
Intervention Model Description: a group of normal hearing and hearing-impaired participants
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental: normal-hearing and hearing-impaired participants (Experimental): normal and hearing-impaired participants
  Interventions: Procedure: Effect of several processing on the auditory distance perception

INTERVENTIONS:
Procedure: Effect of several processing on the auditory distance perception — The focus is a comparison of hearing instrument algorithms on the auditory distance perception

SUMMARY:
A methodical evaluation of novel sound changing principles in CE-labelled Sonova brand hearing instruments (e.g. Phonak hearing instruments) is intended to be conducted on hearing impaired participants. These sound changing principles are enabled by respective hearing instrument technologies and hearing instrument algorithms. The aim of the study is to investigate and assess strengths and weaknesses of these novel sound changing principles in terms of hearing performance to determine their application in hearing instruments (Phase of development). Both, objective laboratory measurements as well as subjective evaluations in real life environment will be carried out. This will be a controlled, single blinded and randomised active comparator clinical evaluation which will be conducted mono centric at the University Hospital of Zürich.

ELIGIBILITY:
Participants fulfilling any of the following inclusion criteria are eligible for the study:

* Adult persons (minimum age: 18 years)
* Healthy outer ear (without previous surgical procedures, except cochlear implantation)
* Ability to fill in a questionnaire conscientiously
* Informed Consent as documented by signature

Normal hearing participants

• Adult persons with audiometric normal hearing thresholds

Hearing impaired participants

* Adult hearing impaired persons with and without (experience with) hearing aids
* Adult hearing impaired persons with cochlear implant(s)

The presence of any one of the following exclusion criteria will lead to exclusion of the participant:

* Contraindications to the MD in this study, e.g. known hypersensitivity or allergy to the investigational product
* Limited mobility and not in the position to attend weekly appointments
* Limited ability to describe listening impressions/experiences and the use of the hearing aid
* Inability to produce a reliable hearing test result
* Massively limited dexterity
* Known psychological problems
* Known central hearing disorders

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2019-11-18 (Actual); Primary Completion 2020-01-31 (Actual); Study Completion 2020-01-31 (Actual)

PRIMARY OUTCOMES:
Success rate of the distance discrimination | 8 weeks
  Participants are asked whether an audio stimulus is closer or further at the end of the stimulus than at its beginning. The success rate is measured as a function of the test conditions.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Zurich, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gatehouse S, Noble W. The Speech, Spatial and Qualities of Hearing Scale (SSQ). Int J Audiol. 2004 Feb;43(2):85-99. doi: 10.1080/14992020400050014. PMID 15035561
- [Background] Mueller MF, Meisenbacher K, Lai WK, Dillier N. Sound localization with bilateral cochlear implants in noise: how much do head movements contribute to localization? Cochlear Implants Int. 2014 Jan;15(1):36-42. doi: 10.1179/1754762813Y.0000000040. Epub 2013 Nov 25. PMID 23684420
- [Background] Catic J, Santurette S, Dau T. The role of reverberation-related binaural cues in the externalization of speech. J Acoust Soc Am. 2015 Aug;138(2):1154-67. doi: 10.1121/1.4928132. PMID 26328729
- [Background] Simon LS, Zacharov N, Katz BF. Perceptual attributes for the comparison of head-related transfer functions. J Acoust Soc Am. 2016 Nov;140(5):3623. doi: 10.1121/1.4966115. PMID 27908072
- See also: Link the the previous part of the study — https://clinicaltrials.gov/ct2/show/NCT03774030?term=sonova&draw=4&rank=26